CLINICAL TRIAL: NCT07386054
Title: The Effectiveness of Binaural Beats on Midazolam Requirement During Cesarean Section With Spinal Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2025-0594
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy, Cesarean Section, Spinal Anesthesia
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ear phone with binaural beats (Experimental): Patient group who receives remimazolam for sedation after delivery
  Interventions: Biological: binaural beats
- ear phone with no sound (Active Comparator): Patient group who receives midazolam for sedation after delivery
  Interventions: Biological: Midazolam

INTERVENTIONS:
Biological: binaural beats — Immediately after admission to the operating room, patients will be fitted with earphones connected to an audio device (Sony Digital Media Player, NW-A306), and the assigned auditory intervention will be initiated. Patients allocated to the binaural beats group will receive auditory stimuli through the earphones, with a frequency difference of 0.5-4 Hz between the two ears to generate an interference frequency via binaural beats. No background music will be provided, and the volume will be set at a level comparable to normal conversational speech.
  Arms: ear phone with binaural beats
Biological: Midazolam — Patients in the control group will wear the earphones without exposure to any auditory stimuli.
  Arms: ear phone with no sound

SUMMARY:
Spinal anesthesia is preferred for cesarean section in many institutions due to concerns regarding the potential effects of general anesthetic agents on the fetus. However, during cesarean section under spinal anesthesia, parturients remain fully conscious and may experience significant anxiety, tension, or fear intraoperatively. For this reason, sedative agents such as midazolam are commonly administered after delivery, once the risk of neonatal exposure is considered minimal, to facilitate maternal sedation. Nevertheless, administration of midazolam at higher doses may be associated with adverse maternal effects, including respiratory depression, apnea, and hemodynamic instability.

Binaural beats are a brainwave entrainment technique in which two auditory stimuli of slightly different frequencies are presented separately to each ear, resulting in the perception of an interference frequency that may induce synchronization of brain activity. Previous studies have reported that exposure to binaural beats designed to generate low-frequency brainwaves associated with relaxation or sleep may reduce pain, anxiety, and promote sedation in both adult and pediatric populations.

The investigators hypothesize that the use of binaural beats during cesarean section under spinal anesthesia may reduce the required dose of midazolam for sedation, thereby decreasing the risk of drug-related adverse effects. The primary objective of this study is to evaluate whether exposure to binaural beats reduces the total dose of midazolam required for sedation in parturients undergoing cesarean section under spinal anesthesia. Secondary objectives include comparison of perioperative anxiety levels, maternal satisfaction, and other perioperative outcomes between the binaural beats group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥20 years undergoing cesarean section under spinal anesthesia who request intraoperative sedation.

Exclusion Criteria:

A. Parturients with hearing impairment or those using hearing aids B. Parturients who have received opioid analgesics or sedative medications within 1 week prior to enrollment C. Parturients with known hypersensitivity to benzodiazepines D. Parturients in whom a difficult airway is anticipated E. Parturients with arrhythmias, cardiovascular disease, impaired cardiac function, or reduced circulating blood volume F. Parturients with severe respiratory disease for whom the use of sedative medications is considered inappropriate G. Parturients with hepatic failure H. Parturients with renal failure or those receiving dialysis I. Parturients with other significant maternal medical histories or fetal conditions (e.g., fetal anomalies, intrauterine growth restriction) that are considered likely to increase maternal anxiety J. Patients who are unable to read the informed consent form (e.g., foreign nationals) K. Participants deemed inappropriate for participation in this clinical trial at the discretion of the investigator or study personnel

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — As this study evaluates the dose of midazolam administered from the initiation of sedation until achievement of an Observer's Assessment of Alertness/Sedation (OAA/S) score of ≤3 during cesarean section,, only female participants are eligible to this study.
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
the total dose of midazolam administered to achieve a score of ≤3 on the Observer's Assessment of Alertness/Sedation (OAA/S) scale during sedation induction. | 1, 2, 3, 4, 5, 10, 20, 30 minutes after sedative administration
  The cumulative dose of midazolam administered from the initiation of sedation until achievement of an OAA/S score of ≤3 will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Hyun Kim, Professor, Principal Investigator — Severance Hospital

IPD SHARING:
Plan to Share IPD: No